CLINICAL TRIAL: NCT04968925
Title: Evaluation of Comfort for Two Marketed Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6456
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- O1D/P1 (Experimental): Eligible subjects that are habitual wearers of daily disposable soft contact lenses will randomly be assigned sequence (O1D/P1)
  Interventions: Device: ACUVUE Oasys 1-Day; Device: Precision 1
- P1/O1D (Experimental): Eligible subjects that are habitual wearers of daily disposable soft contact lenses will randomly be assigned sequence (P1/O1D)
  Interventions: Device: ACUVUE Oasys 1-Day; Device: Precision 1

INTERVENTIONS:
Device: ACUVUE Oasys 1-Day — TEST
Device: Precision 1 — CONTROL

SUMMARY:
This study is a 2-phase adaptive approach utilizing a 2×2 crossover design. The study lenses will be worn in a bilateral fashion for a period of approximately 1-week each.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 40 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft spherical contact lenses in both eyes in a daily disposable wear modality. Habitual wear is defined as a minimum of 8 hours of wear per day, for a minimum of 4 days per week during the past 4 weeks.
5. By self-report, typically uses computer screens and other digital devices (phones, tablets) at least 30 hours per week.
6. The vertex-corrected best spherical distance refraction (rounded to nearest 0.25 D) must be between -1.00 and -4.00 DS (inclusive) in each eye.
7. The magnitude of the cylinder component of the subject's distance refraction must be 1.00 DC or less.
8. The subject must have best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or breastfeeding
2. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See Section 9.1 for additional details regarding excluded systemic medications.
3. Have had any previous ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, cataract, etc.).
4. Habitually wear monovision, multifocal, toric, or extended wear contact lens correction
5. Have participated in any contact lens or lens care product clinical trial within 14 days prior to study enrollment
6. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician)
7. Have a history of amblyopia or strabismus.
8. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (eg, SynergEyes) within the past 6 months.
9. Have clinically significant (Grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
10. Have any ocular infection.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 302 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (10):
- United States (10):
  - James R. Dugue Optometry, Mission Viejo, California
  - Maitland Vision Center, Maitland, Florida
  - Flora Chen Poveda, OD, PA, Orange Park, Florida
  - Visual Eyes, Inc, Roswell, Georgia
  - VisionPoint Center, Bloomington, Illinois
  - ABQ Eye Care, Albuquerque, New Mexico
  - ProCare Vision Center, Granville, Ohio
  - Optometry Group LLC, Memphis, Tennessee
  - Gulf Coast Vision Center, Inc., Houston, Texas
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-Phase study. In Phase I, 75 subjects were enrolled. Of those enrolled into Phase I, all subjects were dispensed at least 1 study lens. Of those dispensed, 72 completed Phase I, while 3 subject discontinued. In Phase II, 227 subjects were enrolled. Of those enrolled, all subjects were dispensed at least 1 study lens. Of those dispensed in Phase II 206 completed the Phase II, while 21 subjects discontinued from Phase II.
Pre-assignment Details: Phase I and Phase II are mutually exclusive. Data collected from Phase I was used to estimate the sample size requirements for Phase II primary endpoints.
Groups:
- Senofilcon A (C3)/Verofilcon A (Phase I); Senofilcon A (C3)/Verofilcon A (Phase II): Subjects randomized to this sequence received the senofilcon A (C3) lens during the first period and then received the verofilcon A lens during the second period.
- Verofilcon A/ Senofilcon A (C3) (Phase I): verofilcon A/ senofilcon A (C3) (Phase I) Subjects randomized to this sequence received the verofilcon A lens during the first period and then received the senofilcon A (C3) lens during the second period.
- Verofilcon A/ Senofilcon A (C3) (Phase II): Subjects randomized to this sequence received the verofilcon A lens during the first period and then received the senofilcon A (C3) lens during the second period.
Period: Phase I- Period 1
Arm/Group | Senofilcon A (C3)/Verofilcon A (Phase I) | Verofilcon A/ Senofilcon A (C3) (Phase I) | Senofilcon A (C3)/Verofilcon A (Phase II) | Verofilcon A/ Senofilcon A (C3) (Phase II)
Started | 35 | 40 | 0 | 0
Completed | 34 | 38 | 0 | 0
Not Completed | 1 | 2 | 0 | 0
Not completed — COVID-19 related | 0 | 1 | 0 | 0
Not completed — Subject enrolled in error | 1 | 1 | 0 | 0
Period: Phase I- Period 2
Arm/Group | Senofilcon A (C3)/Verofilcon A (Phase I) | Verofilcon A/ Senofilcon A (C3) (Phase I) | Senofilcon A (C3)/Verofilcon A (Phase II) | Verofilcon A/ Senofilcon A (C3) (Phase II)
Started | 34 | 38 | 0 | 0
Completed | 34 | 38 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase II- Period 1
Arm/Group | Senofilcon A (C3)/Verofilcon A (Phase I) | Verofilcon A/ Senofilcon A (C3) (Phase I) | Senofilcon A (C3)/Verofilcon A (Phase II) | Verofilcon A/ Senofilcon A (C3) (Phase II)
Started | 0 | 0 | 112 | 115
Completed | 0 | 0 | 105 | 109
Not Completed | 0 | 0 | 7 | 6
Not completed — COVID-19 Related | 0 | 0 | 6 | 6
Not completed — Subject enrolled in error | 0 | 0 | 1 | 0
Period: Phase II -Period 2
Arm/Group | Senofilcon A (C3)/Verofilcon A (Phase I) | Verofilcon A/ Senofilcon A (C3) (Phase I) | Senofilcon A (C3)/Verofilcon A (Phase II) | Verofilcon A/ Senofilcon A (C3) (Phase II)
Started | 0 | 0 | 105 | 109
Completed | 0 | 0 | 101 | 105
Not Completed | 0 | 0 | 4 | 4
Not completed — COVID-19 related | 0 | 0 | 4 | 3
Not completed — Incorrectly dispensed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Phase I: All subjects that were enrolled into Phase I of the study.
- Phase II: All subjects that were enrolled in Phase II of the study
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 75 | 227 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.4 (6.94) | 29.4 (6.23) | 29.2 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 172 | 222
  Male | 25 | 55 | 80
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 6 | 7 | 13
  American Indian or Alaska Native | 0 | 4 | 4
  Black or African American | 6 | 24 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 63 | 191 | 254
Region of Enrollment [Number; unit: Participants]
  United States | 75 | 227 | 302

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort (Phase I)
Description: Overall Comfort was assessed using the individual questionnaire item "How would you rate the study contact lenses on: Overall Comfort" with a 6-point Excellence Response Set of 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All Subjects that completed Phase I of the study without a major protocol deviation impacting a primary endpoint.
Measure: Number; unit: Number of responses
Groups:
- Senofilcon A (C3): Subjects that wore the senofilcon A (C3) lens in either the first or second period of Phase I study.
- Verofilcon A: Subjects that wore the verofilcon A lens in either the first or second period of Phase I study.
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 72 | 72
Number of responses
  Excellent | 45 | 32
  Very Good | 20 | 23
  Good | 5 | 9
  Fair | 2 | 7
  Poor | 0 | 1
Statistical Analysis 1: Comparison: Senofilcon A (C3) vs Verofilcon A; Phase I was not powered to test for non-inferiority for any endpoints. The data collected from this Phase was used to estimate the sample size required to achieve the primary endpoints for Phase II of the study; Test type: Non-Inferiority — A non-inferiority margin of 10% was used; Generalized linear Mixed Model Analysis; Odds Ratio (OR) = 4.24, 95% CI 2-sided [0.80 to 22.54] — Odds ratio was calculated as Test over Control

2. Primary Outcome: End of Day Comfort (Phase I)
Description: End of day Comfort was assessed using the individual questionnaire item "How would you rate the study contact lenses on: comfort at the end of the day" with aa 6-point Excellence Response Set of 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All Subjects that completed Phase I of the study without a major protocol deviation impacting a primary endpoint.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 72 | 72
Number of responses
  Excellent | 29 | 25
  Very Good | 28 | 17
  Good | 9 | 16
  Fair | 4 | 10
  Poor | 2 | 4
Statistical Analysis 1: Comparison: Senofilcon A (C3) vs Verofilcon A; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — A non-inferiority margin of 10% was used; Generalized linear Mixed Model Analysis; Odds Ratio (OR) = 3.44, 95% CI 2-sided [1.16 to 10.16] — Odds ratio was calculated as Test over Control

3. Primary Outcome: End of Day Dryness (Phase I)
Description: End of day Dryness was assessed using the individual questionnaire item "How would you rate the study contact lenses on: Keeping your eyes from feeling dry at the end of the day" with a 6-point Excellence Response Set of 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All Subjects that completed Phase I of the study without a major protocol deviation impacting a primary endpoint.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 72 | 72
Number of responses
  Excellent | 26 | 22
  Very Good | 28 | 20
  Good | 9 | 12
  Fair | 6 | 12
  Poor | 3 | 6
Statistical Analysis 1: Comparison: Senofilcon A (C3) vs Verofilcon A; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — A non-inferiority margin of 10% was used; Generalized linear Mixed Model Analysis; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.05 to 6.76] — Odds ratio was calculated as Test over Control

4. Primary Outcome: End of Day Comfort (Phase II)
Description: End of day Comfort was assessed using the individual questionnaire item "How would you rate the study contact lenses on: comfort at the end of the day" with a 6-point Excellence Response Set of 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Groups:
- Senofilcon A (C3): Subjects that wore the senofilcon A (C3) lens in either the first or second period of Phase II study.
- Verofilcon A: Subjects that wore the verofilcon A lens in either the first or second period of Phase II study.
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Excellent | 89 | 65
  Very Good | 63 | 59
  Good | 24 | 39
  Fair | 26 | 34
  Poor | 8 | 13
Statistical Analysis 1: Comparison: Senofilcon A (C3) vs Verofilcon A; It was calculated based on Phase I using Stroup's Method that 200 subjects were required to test superiority for each endpoint in Phase II; Test type: Superiority — The Fallback Method was used to test primary hypotheses in Phase II. An alpha of 0.167 was allocated for each test. Every successful test passed the "unused" alpha to the next; Generalized linear Mixed Model Analysis; Odds Ratio (OR) = 1.76, 98.33% CI 2-sided [1.09 to 2.83] — Odds ratio was calculated as Test over Control

5. Primary Outcome: End of Day Dryness (Phase II)
Description: as for outcome 3
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Excellent | 83 | 53
  Very Good | 55 | 64
  Good | 27 | 32
  Fair | 32 | 41
  Poor | 13 | 20
Statistical Analysis 1: Comparison: Senofilcon A (C3) vs Verofilcon A; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Generalized linear Mixed Model Analysis; Odds Ratio (OR) = 1.52, 96.66% CI 2-sided [1.02 to 2.28] — Odds ratio was calculated as Test over Control

6. Primary Outcome: Overall Comfort (Phase II)
Description: as for outcome 1
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Excellent | 127 | 104
  Very Good | 44 | 59
  Good | 28 | 30
  Fair | 11 | 13
  Poor | 0 | 3
  Not Applicable | 0 | 1
Statistical Analysis 1: Comparison: Senofilcon A (C3) vs Verofilcon A; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Generalized linear Mixed Model Analysis; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.77 to 2.03] — Odds ratio was calculated as Test over Control

7. Secondary Outcome: Comfort Throughout the Day (Phase II)
Description: Comfort Throughout the Day was assessed using the individual questionnaire item "How would you rate the study contact lenses on: Keeping your eyes feeling comfortable from morning to night" with a 6-point Excellence Response Set of 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Excellent | 96 | 76
  Very Good | 55 | 56
  Good | 29 | 45
  Fair | 26 | 25
  Poor | 4 | 8

8. Secondary Outcome: Comfort While Using Digital Devices (Phase II)
Description: Comfort while Using Digital Devices was assessed using the individual questionnaire item "How would you rate the study contact lenses on: Remaining comfortable while using computer screens and other digital devices (phones, tablets)" with a 6-point Excellence Response Set of 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Not Applicable | 1 | 2
  Excellent | 111 | 90
  Very Good | 46 | 61
  Good | 33 | 31
  Fair | 17 | 22
  Poor | 2 | 4

9. Secondary Outcome: Dryness While Using Digital Devices (Phase II)
Description: Dryness while using Digital Devices was assessed using the individual questionnaire item "How would you rate the study contact lenses on: Keeping your eyes from feeling dry while using computer screens and other digital devices (phones, tablets)." with a 6-point Excellence Response Set of 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Not Applicable | 0 | 2
  Excellent | 102 | 79
  Very Good | 55 | 63
  Good | 25 | 31
  Fair | 22 | 31
  Poor | 6 | 4

10. Secondary Outcome: Lens Awareness Upon Insertion (Phase II)
Description: Lens Awareness Upon Insertion was assessed using the individual questionnaire item "I lost awareness of these lenses shortly after inserting them (within one minute)" with a 5-point Agreement Response Set of 1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree and 5: Strongly Agree. Subject responses are reported by lens using frequencies.
Time Frame: 1-Minute Post lens fitting
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 220 | 221
Number of responses
  Strongly Disagree | 16 | 16
  Disagree | 6 | 13
  Neither Agree nor Disagree | 7 | 8
  Agree | 65 | 71
  Strongly Agree | 126 | 113

11. Secondary Outcome: Comfort Upon Insertion (Phase II)
Description: Comfort Upon Insertion was assessed using the individual questionnaire item "These lenses were comfortable shortly after inserting them (within one minute)" with a 5-point Agreement Response Set of 1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree and 5: Strongly Agree. Subject responses are reported by lens using frequencies.
Time Frame: 1-Minute Post lens fitting
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 220 | 221
Number of responses
  Strongly Disagree | 2 | 6
  Disagree | 0 | 3
  Neither Agree nor Disagree | 4 | 9
  Agree | 61 | 64
  Strongly Agree | 153 | 139

12. Secondary Outcome: Overall Ease of Handling (Phase II)
Description: Overall Ease of Handling was assessed using the individual questionnaire item "How would you rate the study contact lenses on: Overall ease of handling the lenses (putting them on and taking them off)." with a 6-point Excellence Response Set of 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Not Applicable | 0 | 2
  Excellent | 140 | 112
  Very Good | 36 | 40
  Good | 23 | 32
  Fair | 11 | 16
  Poor | 0 | 8

13. Secondary Outcome: Ease of Insertion (Phase II)
Description: Ease of Insertion was assessed using the individual questionnaire item "How would you rate the study contact lenses on: Ease of putting the lenses on your eyes " with a 6-point Excellence Response Set of 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Not Applicable | 0 | 2
  Excellent | 145 | 136
  Very Good | 39 | 36
  Good | 20 | 26
  Fair | 6 | 8
  Poor | 0 | 2

14. Secondary Outcome: Ease of Removal (Phase II)
Description: Ease of Removal was assessed using the individual questionnaire item "how would you rate the study contact lenses on: Ease of taking the lenses off your eyes" with a 6-point Excellence Response Set of 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Subject responses are reported by lens using frequencies.
Time Frame: 1-Week Follow-up
Population: All subjects dispensed a study lens in Phase II with 1-week follow-up data for both study lenses.
Measure: Number; unit: Number of responses
Arm/Group | Senofilcon A (C3) | Verofilcon A
Number analyzed (Participants) | 210 | 210
Number of responses
  Not Applicable | 0 | 3
  Excellent | 139 | 100
  Very Good | 37 | 41
  Good | 22 | 30
  Fair | 11 | 21
  Poor | 1 | 15

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Study duration for Phase I and Phase II were approximately 3-weeks per subject.
Groups:
- Phase I -Senofilcon A (C3): Subjects that wore the senofilcon A (C3) lens in either the first or second period during Phase I of the study.
- Phase I -Verofilcon A: Subjects that wore the verofilcon A lens in either the first or second period during Phase I of the study.
- Phase II -Senofilcon A (C3): Subjects that wore the senofilcon A (C3) lens in either the first or second period during Phase II of the study.
- Phase II -Verofilcon A: Subjects that wore the verofilcon A lens in either the first or second period during Phase II of the study.
Arm/Group | Phase I -Senofilcon A (C3) | Phase I -Verofilcon A | Phase II -Senofilcon A (C3) | Phase II -Verofilcon A
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/74 | 0/221 | 0/220
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/74 | 0/221 | 0/220
Other Adverse Events (participants affected / at risk) | 0/73 | 0/74 | 0/221 | 0/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04968925/Prot_SAP_000.pdf